CLINICAL TRIAL: NCT03544853
Title: Computational Design, Fabrication, and Evaluation of Optimized Patient-Specific Transtibial Prosthetic Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1101004280; R01EB024531-01 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-06-04 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Amputation Stump
Keywords: Prosthetic socket; Biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prosthetic socket evaluation (Experimental): Intervention: Prosthetic socket for transtibial amputee. A subject's conventional prosthetic socket is compared to a novel prosthetic socket designed as part of the research. For standing and walking exercises the following will be assessed. 1) local skin contact pressures, 2) metabolic power, 3) gait parameters (symmetry indices for joint angles, positions, torques, and also ground reaction forces), and 4) the socket evaluation questionnaire.
  Interventions: Device: Prosthetic socket for transtibial amputee

INTERVENTIONS:
Device: Prosthetic socket for transtibial amputee — To wear a prosthetic socket for evaluation of comfort and biomechanical metrics such as skin loading conditions.

SUMMARY:
The overall goal of this study is to further develop and clinically assess a computational and data-driven design and manufacturing framework for mechanical interfaces that quantitatively produces transtibial prosthetic sockets in a faster and more cost-effective way than conventional processes. The main hypothesis of this proposal is that the novel quantitative interface is equivalent to, or better than, a conventional interface in terms of: 1) gait symmetry, 2) skin contact pressures, 3) skin surface temperature, and 4) comfort as evaluated from a questionnaire.

DETAILED DESCRIPTION:
Title: Computational Design, Fabrication, and Evaluation of Optimized Patient-Specific Transtibial Prosthetic Sockets

Principle Investigator: Dr. Hugh Herr

Background: The overall goal of this application is to further develop and clinically assess a computational and data-driven design and manufacturing framework for mechanical interfaces that quantitatively produces transtibial prosthetic sockets in a faster and more cost-effective way than conventional processes. Traditionally, prosthetic socket production has been a craft activity, based primarily on the experience of the prosthetist. Even with advances in computer-aided design and computer-aided manufacturing (CAD/CAM), the design process remains manual. The manual nature of the process means it is non-repeatable and currently largely non-data-driven, and quantitative data is either not obtained or insufficiently employed. Furthermore, discomfort, skin problems and pressure ulcer formation remain prevalent. Through the proposed computational modeling framework, a repeatable, data-driven and patient-specific design process is made available which is based on scientific rationale.

Objective/hypothesis: The main hypothesis of this proposal is that a socket, designed using the novel computational design framework, is equivalent to, or better than, a conventional socket (designed by a prosthetist) in terms of: 1) gait symmetry, 2) skin contact pressures, 3) skin surface temperature, and 4) comfort as evaluated from a questionnaire. Our hypothesis is supported by the presented pilot data which shows reduced or equivalent skin contact pressures and subject reported comfort levels for several critical anatomical regions.

Specific Aims: 1) Subject-specific biomechanical modeling for N=18 subjects, 2) Computational design and fabrication of sockets for N=18 subjects, and 3) Clinical evaluation of novel sockets for N=18 subjects.

Study Design: A cohort of 18 subjects will be recruited for this study. MRI or CT data will be recorded for all subjects. Through image segmentation geometrically accurate 3D finite element analysis (FEA) models will be constructed. The resulting predictive FEA models will then be used in a novel, data-driven, and automated computational design framework for prosthetic sockets, to design prosthetic sockets for all subjects. The framework optimizes the socket designs, as assessed by skin contact pressures and internal tissue strain, through iterative adjustment of the virtual tests sockets. Final designs are subsequently 3D printed. To evaluate the prosthetic sockets with each of the subjects each subject will do a standing and walking exercise using their conventional sockets or the novel sockets. Meanwhile skin contact pressures and temperatures are recorded, gait symmetry data is collecetd, and socket comfort is assessed using a questionnaire. Together this data provides a quantitative and qualitative evaluation and comparison of the novel and conventional sockets.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 years old
* Amputation type: Transtibial amputation (bilateral or unilateral) which took place >1 year prior to study
* Activity or K-level: At least K3
* Socket quality: The subject's conventional socket(s) should be deemed of high quality and comfortable
* MRI safety: Subjects should be able to undergo MRI

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Local skin pressure while wearing a socket | Assessed once during (clinical) socket comfort evaluation phase. Measurements are for standing and walking exercises for the conventional and novel socket.
  Local skin contact pressures (in Newton per square meter) are assessed using pressure sensors positioned on the skin surface. Local pressures relate to comfort which is the topic of investigation. These measurements are performed during the (clinical) socket comfort evaluation phase which is typically 3 months after the initial data acquisition phase for each subject. Measurements take place once and in a single session. As such only a single time point is investigated (the time point of the experiment is not a relevant or investigated parameter). The data is compared across subjects and socket types.
Skin surface temperature difference | Assessed once during (clinical) socket comfort evaluation phase. Measurements are for standing and walking exercises for the conventional and novel socket.
  Skin surface temperatures (in Celsius) are assessed using a Flir thermal camera, with images taken immediately post-kinematic walking trial. From these measurements the average residuum skin surface temperature is assessed for 4 different view directions: anterior, posterior, medial, and lateral. Measurements take place once and in a single session. As such only a single time point is investigated (the time point of the experiment is not a relevant or investigated parameter). The data is compared across subjects and socket types.
Gait parameter asymmetry | Assessed once during (clinical) socket comfort evaluation phase. Measurements are for standing and walking exercises for the conventional and novel socket.
  Socket fit (and discomfort) influences musculoskeletal behavior and may alter gait patterns. Subjects are equipped with markers tracked (units of mm) using a motion capture system (T40s, Vicon Motion Systems Ltd, Oxford, UK). Ground reaction forces (units Newton) are also recorded. From these measurements gait symmetry indices for: joint angles, positions, torques, and ground reaction forces, are computed. These measurements are performed during the (clinical) socket comfort evaluation phase which is typically 3 months after the initial data acquisition phase for each subject. Measurements take place once and in a single session. As such only a single time point is investigated (the time point of the experiment is not a relevant or investigated parameter). The data is compared across subjects and socket types.
Socket evaluation questionnaire | Assessed once during (clinical) socket comfort evaluation phase. Measurements are for sitting, standing and walking exercises for the conventional and novel socket.
  Socket fit and discomfort is assessed using a questionnaire created to document patient experiences and preferences while using prosthetic interfaces (liners, sockets) both over a longitudinal timeline and on an immediate basis. After establishing subject baselines for socket use, patients complete a section that instructs them to evaluate the novel prosthetic socket provided against their conventional prosthetic socket. Subjects complete the questionnaire via a HIPAA compliant surveying instrument on Redcap, and questions are tailored to minimize bias through adoption of verified metrics (such as those from the TAPES-R instrument) or by the use of sliding scales that eliminate the need for constrained integer number input. The data is analyzed by subject, across subjects as a whole, and socket types.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh M Herr, PhD, Principal Investigator — Massachusetts Institute of Technology, Media Lab
Locations (2):
- Massachusetts Institute of Technology, Media Lab, Cambridge, Massachusetts, United States
- Tecnologico de Monterrey, Biomechatronics Lab, Nuevo México, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03544853/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03544853/SAP_001.pdf
  • Informed Consent Form (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03544853/ICF_002.pdf